CLINICAL TRIAL: NCT03350828
Title: The CHEC-SC Cohort Study: CHaractErizing CFTR Modulated Changes in Sweat Chloride and Their Association With Clinical Outcomes
Brief Title: CHaractErizing CFTR Modulated Changes in Sweat Chloride and Their Association With Clinical Outcomes
Acronym: CHEC-SC
Status: Active, not recruiting | Type: Observational
Sponsor: Nicole Hamblett (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Nicole Hamblett, Professor in the Department of Pediatrics in the Division of Pulmonary Medicine, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Other Study IDs: CHEC-OB-17
Record Dates: First submitted 2017-11-09; First posted 2017-11-22 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
Keywords: CF; Cystic Fibrosis; Sweat; Sweat chloride; CFTR Modulator
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a multicenter, cross-sectional, cohort study which will collect contemporary sweat chloride (SC) values from approximately 5000 Cystic Fibrosis (CF) patients prescribed and currently receiving commercially approved Cystic Fibrosis transmembrane conductance regulator (CFTR) modulator therapies.

DETAILED DESCRIPTION:
Eligible subjects who have been prescribed and chronically taking a commercially approved CFTR modulator for at least 3 months will be enrolled for a single visit to collect sweat to be analyzed for SC at their local site laboratory. Limited clinical data obtained at this visit will be augmented by retrospective and prospective data obtained from the Cystic Fibrosis Foundation Patient Registry (CFFPR). Study subjects who have been prescribed and switch to an alternative commercially approved CFTR modulator will be approached to re-enroll in the study after being on the alternative modulator for at least 3 months so that a new SC value can be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative
2. Enrolled in the CFFPR
3. Male or female ≥ 4 months of age on day of study visit
4. Diagnosis of CF.
5. Current treatment with a prescribed commercially approved CFTR modulator for at least 90 days prior to enrollment
6. Able to perform the testing and procedures required for this study, as judged by the investigator

Additional Inclusion Criteria for CHEC-PKPD Sub-Study:

1. Male or female ≥ 6 years of age on day of study visit.
2. Current treatment with elexacaftor/tezacaftor/ivacaftor for at least 90 days prior to enrollment.
3. Last dose of elexacaftor/tezacaftor/ivacaftor taken at least 24hours and last dose of ivacaftor taken at least 12 hours prior to trough blood draw on day of visit.

Exclusion Criteria:

1. Presence of a condition or abnormality that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data
2. Currently enrolled in an investigational trial (including open-label follow-on studies and Early Access Programs (EAP) of an agent expected to have an impact on sweat chloride (refer to current list provided on study website)

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cystic Fibrosis Care Centers
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
mean change in sweat chloride pre- to post- modulator therapy | through study completion, an average of 1 year
  mean change in sweat chloride pre- to post- modulator therapy

CONTACTS AND LOCATIONS:
Overall Officials: Edith Zemanick, MD, Principal Investigator — University of Colorado, Denver; Michael Konstan, MD, Principal Investigator — Case Western Reserve University; Nicole Mayer-Hamblett, PhD, Principal Investigator — Seattle Children's Hospital
Locations (52):
- United States (52):
  - The Children's Hospital Alabama, University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego, La Jolla, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - The Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Children's Healthcare of Atlanta and Emory University, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Michigan Medicine, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - SSM Health Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Cystic Fibrosis Center of Western New York, Buffalo, New York
  - New York Medical College at Westchester Medical Center, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Hershey Medical Center Pennsylvania State University, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee CF Care and Research Center, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Texas Southwestern / Children's Health, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Primary Children's Cystic Fibrosis Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - West Virginia University - Morgantown, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] VanDevanter DR, Zemanick ET, Konstan MW, Ren CL, Odem-Davis K, Emerman I, Young J, Mayer-Hamblett N; CHEC-SC Study Group. Willingness of people with cystic fibrosis receiving elexacaftor/tezacaftor/ivacaftor (ETI) to participate in randomized modulator and inhaled antimicrobial clinical trials. J Cyst Fibros. 2023 Jul;22(4):652-655. doi: 10.1016/j.jcf.2023.04.007. Epub 2023 Apr 24. PMID 37100705